CLINICAL TRIAL: NCT07008469
Title: A Global Phase 3 Open-Label Extension Study to Assess the Long-Term Safety, Tolerability, and Efficacy of Intravenous AOC 1001 for the Treatment of Myotonic Dystrophy Type 1
Brief Title: Global Open-Label Extension Study of Del-desiran for the Treatment of DM1
Acronym: HARBOR-OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOC 1001-CS4
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Myotonic Dystrophy Type 1; DM1; Myotonic Dystrophy; Myotonia; Myotonic Dystrophy 1; Myotonic Disorders; Steinert Myotonic Dystrophy; Steinert Disease
Keywords: DM1; Myotonic Dystrophy; Myotonic Dystrophy 1; Myotonia; Myotonic Dystrophy Type 1 (DM1); Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Steinert; Myotonic Muscular Dystrophy; HARBOR-OLE; Avidity Biosciences; Avidity; AOC 1001; Del-desiran; Delpacibart etedesiran; HARBOR
MeSH Terms: conditions — Myotonic Dystrophy; Myotonia; Myotonic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Del-desiran (Experimental): Del-desiran (AOC 1001) will be administered seven times per year for up to 4 years.
  Interventions: Drug: Del-desiran (AOC 1001)

INTERVENTIONS:
Drug: Del-desiran (AOC 1001) — Del-desiran will be administered by intravenous (IV) infusion.

SUMMARY:
A Global Phase 3 Open-Label Extension Study to Assess the Long-Term Safety, Tolerability, and Efficacy of Intravenous Delpacibart Etedesiran (abbreviated del-desiran, formerly AOC 1001) for the Treatment of Myotonic Dystrophy Type 1

DETAILED DESCRIPTION:
The study consists of a Screening Period of up to either 4-weeks or 8-weeks depending on the prior parent trial, and up to a 4-year Treatment Period. The anticipated duration is 50 months and 2 weeks (4 years and 2.5 months).

Participants will receive an intravenous infusion of del-desiran at the clinical study site every 8 weeks for a total of 7 doses per year. The final dose will occur at Year 4, Visit 7, followed by a final assessment 8 weeks after the last dose.

An additional subgroup of de novo participants will also be included in a Fixed-Dose PK cohort.

An Independent Data Monitoring Committee (IDMC) comprised of members independent and external to the Sponsor will review safety, tolerability, and efficacy (as needed) data of this study at regular intervals.

ELIGIBILITY:
FROM A PARENT STUDY

Key Inclusion Criteria:

* Completion of any prior AOC 1001 studies with satisfactory completion of dosing and follow-up assessments and satisfactory compliance with the protocol requirements of the parent study, as determined by the Investigator.

Key Exclusion Criteria:

* Breastfeeding, pregnancy, or intent to become pregnant during the study.
* Unwilling to comply with contraceptive requirements.
* Any new conditions or worsening of existing condition that in the opinion of the Investigator would make the participant unsuitable for the study.

FIXED-DOSE PK COHORT

Key Inclusion Criteria:

* Clinical and genetic diagnosis of DM1 and clinically significant hand myotonia.

Key Exclusion Criteria:

* Breastfeeding, pregnancy, or intent to become pregnant during the study
* Unwilling to comply with contraceptive requirements
* Abnormal lab values, conditions or diseases that would make the participant unsuitable for the study
* Diabetes that is not adequately controlled
* History of decompensated heart failure within 3 months of screening. Participants with preexisting pacemaker/ICD are not excluded
* Body Mass Index > 35 kg/m2 at Screening
* Recently treated with an investigational drug or biological agent

Note: Additional protocol defined Inclusion and Exclusion criteria apply

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
TEAEs | From enrollment to the end of treatment at 4 years
  Incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Indiana University (IU), Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- Fondazione Serena Onlus - Centro Clinico NeMO Milano, Milan, Italy
- Japan (2):
  - Aomori Hospital, Aomori, Aomori
  - Osaka University Hospital, Osaka
- Stichting Radboud Universitair Medisch Centrum, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined